CLINICAL TRIAL: NCT06441279
Title: Hyaluronic Acid Versus Platelet Lysate in The Treatment of Temporomandibular Joint Anterior Disc Displacement With Reduction: A Randomized Clinical Trial
Brief Title: Treatment of Tempromandibular Joint Anterior Disc Displacement With Different Materials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0103024OS
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: TMJ Disc Disorder
MeSH Terms: interventions — Injections, Intra-Articular; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): 30 patients that will have intra-articular injection of 2 ml of Platelet lysate (PL).
  Interventions: Procedure: intra-articular injection with Platelet lysate (PL).
- group 2 (Experimental): 30 patients that will have intra-articular injection of Hyaluronic Acid.
  Interventions: Procedure: intra-articular injection with Hyaluronic Acid.

INTERVENTIONS:
Procedure: intra-articular injection with Platelet lysate (PL). — 2 ml of Platelet lysate will be deposited into the superior joint space (SJS) in the affected joint at the entry point slowly
  Arms: group 1
Procedure: intra-articular injection with Hyaluronic Acid. — 2 ml of Hyaluronic Acid will be deposited into the superior joint space (SJS) in the affected joint at the entry point slowly.
  Arms: group 2

SUMMARY:
comparing the clinical efficacy of intra-articular injection of platelet lysate (PL), versus Hyaluronic Acid after arthrocentesis in the management of patients with anterior disc displacement with reduction.

ELIGIBILITY:
Inclusion Criteria:

* Patients that will be diagnosed with anterior disc displacement with reduction (ADDWR) both clinically and through magnetic resonance imaging scan (MRI).
* Patients who will not respond to a previous conservative therapy.
* Patients with pain in temporomandibular joints.
* Patients with normal or limitation in mouth opening.
* Patients with clicking sound.

Exclusion Criteria:

* Patients with previous invasive TMJ surgical procedures.
* Patients with inflammatory or connective tissue diseases.
* Patients with neurologic disorders.
* Patients with history of bony or fibrous adhesion.
* Patients having gross mechanical restrictions and condylar fractures.
* Patients with psychological problems.
* Patients receiving anti-coagulation treatment, non-steroidal anti-inflammatory drugs within 48 hours pre-operatively, corticosteroid injection at the treatment site within one month or systemic use of corticosteroids within 2 weeks.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Maximum inter-incisal opening | 6 months
  Maximum inter-incisal opening will be measured by Vernier caliper and this will be recorded by photographs.

CONTACTS AND LOCATIONS:
Locations (1):
- Heba Elsheikh, Mansoura, Egypt, Egypt